CLINICAL TRIAL: NCT03924063
Title: Safety of the Hemiverse Shoulder Prothesis
Acronym: Hemiverse
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No suitable population available
Sponsor: Balgrist University Hospital (Other)
Collaborators: Salzburger Landeskliniken (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMU27
Record Dates: First submitted 2019-03-26; First posted 2019-04-23 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Rotator Cuff Tear; Hemiarthroplasty
Keywords: total shoulder; failure; salvage
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- conservative treatment (Other): conservative treatment with physical therapy and non steroidal anti-inflammatory drugs
  Interventions: Device: Hemiverse

INTERVENTIONS:
Device: Hemiverse — Implantation of the hemiverse shoulderprothesis

SUMMARY:
This clinical trial investigates the safety and the preliminary clinical benefit of the hemiverse shoulder prosthesis. Implantation of this newly developed hemi-prosthesis is intended for patients who do not qualify for a regular reverse or hemi-prosthesis due to severe medical conditions, poor bone stock or critical status of the rotator cuff. The expected benefit is, that patients will have a minimally invasive surgical procedure, only addressing the humeral shaft, however with the biomechanical advantage of a total reverse shoulder prosthesis, meaning, that with a minimally invasive surgery a comparable result as with a regular total shoulder prosthesis is accomplished. Patients will be closely monitored within the study protocol for 18 months and thereafter in regular interval was as with a normal prosthetic followup.

DETAILED DESCRIPTION:
This clinical trial investigates the safety and the preliminary clinical benefit of the hemiverse shoulder prosthesis. Implantation of this newly developed hemi-prosthesis is intended for patients who do not qualify for a regular reverse or hemi-prosthesis due to severe medical conditions, poor bone stock or critical status of the rotator cuff. To evaluate the clinical condition of the patient a clinical examination with thorough control of the blood parameters (hemoglobin, leucocytes, platelets, infection parameters) and including constant score and the quick dash score will be performed before the operation. To evaluate the bone stock and the musculature a conventional radiological status and a computed tomography of the shoulder will be performed.

Surgical procedure: A delto-pectoral approach is preferred. The incision starts immediately lateral to the coracoid tip and extends to the insertion of the deltoid on the Humerus. The subscapularis tendon is exposed and detached from the humerus. The humeral head is exposed and dislocated from the joint using an oscillating saw the humeral head is resected. The shaft is prepared to receive a regular humeral stem which is definitely implanted with 0° retroversion. A trial implant is inserted and reduced into the joint. Free mobility of the joint is tested and the stability of the implant documented. According to the trial implants the definite implant is assembled and implanted. After reduction of the implant the subscapularis tendon is reattached to the humerus using transosseous sutures. Regular closure of the incision is performed.

After-care:

Immediately post operatively a anteroposterior radiograph is performed. For the first two post-operative weeks the arm is immobilised in a sling and external rotation is allowed until 0° and flexion until 90° in internal rotation. Thereafter gradual increase of active mobility is allowed until the weeks post operatively, when full load bearing of the arm is allowed. Regular followup visits include a constant score, quick dash-score and conventional radiographic status(anteroposterior lateral and axillary view) and are performed to be post-operative 3 months 6 months 1 year and 18 months post operatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥65 years
* Shoulder joint destruction in which known alternatives would constitute either a high patient risk or a high functional failure risk.
* Shoulder destruction suited for hemiarthroplasty except for present cuff failure
* Shoulder destruction for which reverse total shoulder replacement would be a high risk for medical reasons (longer operation, more blood loss) or for advanced glenoid bone destruction
* Written informed consent

Exclusion Criteria:

* Acute or chronic infection Clinical chemistry: C reactive protein <1.5 mg/dl), possible inclusion is under investigator decision.
* Neuroarthropathy
* Moderate to severe motor axillary nerve dysfunction
* Moderate to severe destruction of deltoid muscle
* Fracture of the scapular spine or displaced fracture of the basis of the acromion
* Destruction of more than superior one third of the humeral shaft
* Hematology: hemoglobin (<10 and >16 g/dl), Hematocrit (<36 and >-48%), Anticoagulation
* Poorly controlled diabetes mellitus type I
* Immunosuppressive drugs
* Chronic inflammatory diseases, which the PI estimates contribute to a higher risk of surgery complications
* Inability to cooperate with postoperative regimen or to understand the trial information (dementia)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Safety of implantation of the Hemi verse shoulder prosthesis | Assessments will take place at day 7,
  Adverse Events like fracute, infection, hematoma, nerve demage will be summarized, all clinical data will be evaluated
Safety of implantation of the Hemi verse shoulder prosthesis | Assessments will take place at 6 weeks
  Adverse Events like fracture, dislocation, infection, hematoma, pulmonary embolism, nerve demage will be summarized, all clinical data will be evaluated
Safety of implantation of the Hemi verse shoulder prosthesis | Assessments will take place at 3 months
  Adverse events such as infection stiffness, dislocation, fracture requiring any modification of the expected course and treatment will bed reported at three months.
Safety of implantation of the Hemi verse shoulder prosthesis | Assessments will take place at 6 months
  Adverse Events will be summarized, all clinical data will be evaluated
Safety of implantation of the Hemi verse shoulder prosthesis | Assessments will take place at 12 months
  Adverse Events will be summarized, all clinical data will be evaluated

SECONDARY OUTCOMES:
change of pain using a visual analogue scale: 0-100, 0=no pain 100=maximal imaginable pain | assessment at 6 weeks, 3 months, 6 months and 12 months
  highest pain level within last 25 hours will be recorded on a visual analogue scale
change of active range of motion | assessment at 6 weeks, 3 months, 6 months and 12 months
  active range of motion of the patient will be measured using a handheld goniometer for active elevation, abduction, external rotation and internal rotation
change of strength of abduction | assessment at 6 weeks, 3 months, 6 months and 12 months
  isometric strength of abduction will be measured at 90 degrees scapular abduction using a validated device starting at 3 months postoperatively until end of study

CONTACTS AND LOCATIONS:
Locations (1):
- Landkrankenhaus Salzburg, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No